CLINICAL TRIAL: NCT06421558
Title: Impact of Direct Current Neuromuscular Electrical Stimulation on Physical Therapy Treatment of Lumbosacral Radiculopathy
Brief Title: Impact of Direct Current Electrical Stimulation on Treatment of Lumbosacral Radiculopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NeuFit - Neurological Fitness and Education (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00077736
Record Dates: First submitted 2024-04-08; First posted 2024-05-20 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Radiculopathy Lumbar; Radiculopathy Sacral; Radiculopathy Multiple Sites
Keywords: electrical stimulation; direct current; e-stim; neubie; emg
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Study will be divided into two randomly assigned groups - control and experimental. Control group will receive traditional e-stim treatment with TENS plus physical therapy. Experimental group will receive direct current e-stim treatment with the Neubie device plus physical therapy.
Who Masked: Outcomes Assessor
Masking Description: Outcomes will be assessed by clinicians at Hands on Diagnostics locations. Assessors will be blinded to which intervention participant has received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Neubie Direct Current Electrical Stimulation Device (Experimental): The experimental group subjects follow with 12 sessions of physical therapy over a 6-week period which include 30 min of various physical therapy exercises with the Neubie.
  Interventions: Device: Neubie Direct Current Electrical Stimulation Device
- Transcutaneous Electrical Stimulation (Other): The control group subjects follow with 12 sessions of physical therapy over a 6-week period which include: a 30-min of various physical therapy exercises with TENS application.
  Interventions: Device: Transcutaneous Electrical Stimulation

INTERVENTIONS:
Device: Neubie Direct Current Electrical Stimulation Device — Direct Current Electrical Stimulation Device that uses electrodes non-invasively on the skin to stimulate muscle fibers.
  Arms: Neubie Direct Current Electrical Stimulation Device
Device: Transcutaneous Electrical Stimulation — Transcutaneous Electrical Nerve Stimulation device - uses alternating current delivered through electrodes on the skin.
  Other Names: TENS
  Arms: Transcutaneous Electrical Stimulation

SUMMARY:
This study will compare two methods of electrical stimulation (alternating current and direct current) as an adjunctive therapy to treating lumbosacral radiculopathy. Both types of electrical stimulation have been used in clinical practice for physical therapy, however direct current stimulation is much less common and there is less known about its impact on physical therapy outcomes. The aim of this project is to show the efficacy of a novel device, the Neubie direct current device, compared to traditional TENS unit in clinical physical therapy treatment of radiculopathy. Outcomes measured will include: pain intensity, functional status, neurological status, electrophysiological changes and patient satisfaction.

DETAILED DESCRIPTION:
To determine the efficacy of direct current electrical stimulation (the Neubie device) on long-term symptoms and severity of lumbosacral and thoracic radiculopathy, participants will enroll in a 6-week treatment regimen at one of 16 Hands-On Physical Therapy associated clinic sites listed included in application. The first session will consist of an intake evaluation session that will include: Numeric Pain Scale for pain, Oswestry Disability Index questionnaire to assess functional disability, Straight Leg Raise Test to address nerve root irritation or compression, and Electrophysiological evaluation to determine the nerve function. These tests will serve as baseline (and a within subject control) for the intervention.

Participants will then undergo a specialized radiculopathy protocol that includes traditional PT therapy as well as treatment with the Neubie (or traditional electrical stimulation) both during PT exercises and as additional treatment after sessions. Subjects receive an evaluation session that includes Numeric Pain Scale for pain, Oswestry Disability Index questionnaire to assess functional disability, Straight Leg Raise Test to address nerve root irritation or compression, and Electrophysiological evaluation to determine the nerve function.

The experimental group subjects follow with 12 sessions of physical therapy over a 6-week period which include 30 min of various physical therapy exercises with the Neubie.

The control group subjects follow with 12 sessions of physical therapy over a 6-week period which include: a 30-min of various physical therapy exercises with TENS application.

At the end of the 12 sessions of treatment, subjects receive an evaluation session that includes Numeric Pain Scale for pain, Oswestry Disability Index questionnaire to assess functional disability, Straight Leg Raise Test to address nerve root irritation or compression, Electrophysiological evaluation to determine the nerve function, and a patient satisfaction questionnaire to assess patient satisfaction with the treatment. Participants will receive 12 treatments over 6 weeks. Measurement of these variables will provide both quantitative and qualitative data on the severity of radiculopathy symptoms (see "Tools for data collection" below).

If symptoms of radiculopathy are still present at the 6 week assessment, participants will have the option to continue treatment for up to an additional 12 sessions over 6 more weeks, to a possible maximum of 24 sessions in 12 weeks. Participants will receive a final outcome evaluation session that includes Numeric Pain Rating Scale for pain, Oswestry Disability Index questionnaire to assess functional disability, Straight Leg Raise Test to address nerve root irritation or compression, Electrophysiological evaluation to determine the nerve function, and a patient satisfaction questionnaire to assess patient satisfaction with the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must show evidence of lumbo-sacral radiculopathy as determined by EMG and straight leg raise test.
* Must be able to attend weekly sessions for the 6-week period of the study (no extended travel)
* Must be at least 18 years old.

Exclusion Criteria:

* Currently pregnant
* Cardiac pacemaker
* Active or recent cancer
* Active or recent blood clots
* History of epilepsy
* Open wounds
* Spinal fusion surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
H-Reflex | Pre-intervention
  Electrodes on the skin release tiny electric shocks to stimulate nerves; the amplitude of the nerve signal will be measured for the H-Reflex.
H-Reflex | 6 weeks
  Electrodes on the skin release tiny electric shocks to stimulate nerves; the amplitude of the nerve signal will be measured for the H-Reflex.
H-Reflex | 12 weeks
  Electrodes on the skin release tiny electric shocks to stimulate nerves; the amplitude of the nerve signal will be measured for the H-Reflex.
EMG detection of spontaneous electrical activity | Pre-intervention
  EMG detection of presence of degree of spontaneous electrical activity such as fibrillation potentials and positive sharp waves of muscles innervated by L4, L5, and S1 nerve roots
EMG detection of spontaneous electrical activity | 6 weeks
  EMG detection of presence of degree of spontaneous electrical activity such as fibrillation potentials and positive sharp waves of muscles innervated by L4, L5, and S1 nerve roots
EMG detection of spontaneous electrical activity | 12 weeks
  EMG detection of presence of degree of spontaneous electrical activity such as fibrillation potentials and positive sharp waves of muscles innervated by L4, L5, and S1 nerve roots
Straight Leg Raise Test | Pre-intervention
  Straight Leg Raise Test degrees of movement
Straight Leg Raise Test | 6 weeks
  Straight Leg Raise Test degrees of movement
Straight Leg Raise Test | 12 weeks
  Straight Leg Raise Test degrees of movement
Oswestry Disability Index | Pre-intervention
  Oswestry Disability Index Questionnaire Score
Oswestry Disability Index | 6 weeks
  Oswestry Disability Index Questionnaire Score
Oswestry Disability Index | 12 weeks
  Oswestry Disability Index Questionnaire Score
Numeric Pain Rating Scale | Pre-intervention
  Numeric Pain Rating scale for pain
Numeric Pain Rating Scale | 6 weeks
  Numeric Pain Rating Scale for pain
Numeric Pain Rating Scale | 12 weeks
  Numeric Pain Rating Scale for pain

CONTACTS AND LOCATIONS:
Overall Officials: Ramona von Leden, PhD, Study Director — NeuFit - Neurological Fitness and Education
Locations (15):
- United States (15):
  - NCEPT Physical Therapy, Escondido, California
  - APEX Physical Therapy, Cape Coral, Florida
  - Catalyst Physical Therapy, Clearwater, Florida
  - APEX Physical Therapy, Fort Myers, Florida
  - Kinetix Haile Plantation, Gainesville, Florida
  - Kinetix Arbor Greens - Jonesville, Gainesville, Florida
  - Adams Physical Therapy Services, Portland, Indiana
  - KORT Bardstown, Bardstown, Kentucky
  - KORT Sheperdsville, Shepherdsville, Kentucky
  - Hands On Physical Therpay, Astoria, New York
  - WellHealth Physical Therapy, Deer Park, New York
  - WellHealth Physical Therapy, Hicksville, New York
  - Hands On Physical Therapy of Queens Village, Queens Village, New York
  - Courcier Clinic, Edmond, Oklahoma
  - Spine & Rehab Specialists, El Paso, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berry JA, Elia C, Saini HS, Miulli DE. A Review of Lumbar Radiculopathy, Diagnosis, and Treatment. Cureus. 2019 Oct 17;11(10):e5934. doi: 10.7759/cureus.5934. PMID 31788391
- [Background] Tarulli AW, Raynor EM. Lumbosacral radiculopathy. Neurol Clin. 2007 May;25(2):387-405. doi: 10.1016/j.ncl.2007.01.008. PMID 17445735
- [Background] Sharma H, Lee SW, Cole AA. The management of weakness caused by lumbar and lumbosacral nerve root compression. J Bone Joint Surg Br. 2012 Nov;94(11):1442-7. doi: 10.1302/0301-620X.94B11.29148. PMID 23109619
- [Background] Lewis R, Williams N, Matar HE, Din N, Fitzsimmons D, Phillips C, Jones M, Sutton A, Burton K, Nafees S, Hendry M, Rickard I, Chakraverty R, Wilkinson C. The clinical effectiveness and cost-effectiveness of management strategies for sciatica: systematic review and economic model. Health Technol Assess. 2011 Nov;15(39):1-578. doi: 10.3310/hta15390. No abstract available. PMID 22078311
- [Background] Aono H, Iwasaki M, Ohwada T, Okuda S, Hosono N, Fuji T, Yoshikawa H. Surgical outcome of drop foot caused by degenerative lumbar diseases. Spine (Phila Pa 1976). 2007 Apr 15;32(8):E262-6. doi: 10.1097/01.brs.0000259922.82413.72. PMID 17426622
- [Background] Girardi FP, Cammisa FP Jr, Huang RC, Parvataneni HK, Tsairis P. Improvement of preoperative foot drop after lumbar surgery. J Spinal Disord Tech. 2002 Dec;15(6):490-4. doi: 10.1097/00024720-200212000-00010. PMID 12468976
- [Background] Bauer P, Krewer C, Golaszewski S, Koenig E, Muller F. Functional electrical stimulation-assisted active cycling--therapeutic effects in patients with hemiparesis from 7 days to 6 months after stroke: a randomized controlled pilot study. Arch Phys Med Rehabil. 2015 Feb;96(2):188-96. doi: 10.1016/j.apmr.2014.09.033. Epub 2014 Oct 18. PMID 25449195
- [Background] Glaser JA, Baltz MA, Nietert PJ, Bensen CV. Electrical muscle stimulation as an adjunct to exercise therapy in the treatment of nonacute low back pain: a randomized trial. J Pain. 2001 Oct;2(5):295-300. doi: 10.1054/jpai.2001.25523. PMID 14622808
- [Background] Sluka KA, Walsh D. Transcutaneous electrical nerve stimulation: basic science mechanisms and clinical effectiveness. J Pain. 2003 Apr;4(3):109-21. doi: 10.1054/jpai.2003.434. PMID 14622708
- [Background] Peters EJ, Armstrong DG, Wunderlich RP, Bosma J, Stacpoole-Shea S, Lavery LA. The benefit of electrical stimulation to enhance perfusion in persons with diabetes mellitus. J Foot Ankle Surg. 1998 Sep-Oct;37(5):396-400; discussion 447-8. doi: 10.1016/s1067-2516(98)80048-3. PMID 9798171
- [Background] Gilcreast DM, Stotts NA, Froelicher ES, Baker LL, Moss KM. Effect of electrical stimulation on foot skin perfusion in persons with or at risk for diabetic foot ulcers. Wound Repair Regen. 1998 Sep-Oct;6(5):434-41. doi: 10.1046/j.1524-475x.1998.60505.x. PMID 9844163
- [Background] da Silva MP, Liebano RE, Rodrigues VA, Abla LE, Ferreira LM. Transcutaneous electrical nerve stimulation for pain relief after liposuction: a randomized controlled trial. Aesthetic Plast Surg. 2015 Apr;39(2):262-9. doi: 10.1007/s00266-015-0451-6. Epub 2015 Feb 10. PMID 25665520
- [Background] Ordog GJ. Transcutaneous electrical nerve stimulation versus oral analgesic: a randomized double-blind controlled study in acute traumatic pain. Am J Emerg Med. 1987 Jan;5(1):6-10. doi: 10.1016/0735-6757(87)90281-6. PMID 3545246
- [Background] Zhao M, Bai H, Wang E, Forrester JV, McCaig CD. Electrical stimulation directly induces pre-angiogenic responses in vascular endothelial cells by signaling through VEGF receptors. J Cell Sci. 2004 Jan 26;117(Pt 3):397-405. doi: 10.1242/jcs.00868. Epub 2003 Dec 16. PMID 14679307
- [Background] Kanno S, Oda N, Abe M, Saito S, Hori K, Handa Y, Tabayashi K, Sato Y. Establishment of a simple and practical procedure applicable to therapeutic angiogenesis. Circulation. 1999 May 25;99(20):2682-7. doi: 10.1161/01.cir.99.20.2682. PMID 10338463
- [Background] Thakral G, Kim PJ, LaFontaine J, Menzies R, Najafi B, Lavery LA. Electrical stimulation as an adjunctive treatment of painful and sensory diabetic neuropathy. J Diabetes Sci Technol. 2013 Sep 1;7(5):1202-9. doi: 10.1177/193229681300700510. PMID 24124947
- [Background] Wang TJ, Sung K, Wilburn M, Allbright J. Russian Stimulation/Functional Electrical Stimulation in the Treatment of Foot Drop Resulting from Lumbar Radiculopathy: A Case Series. Innov Clin Neurosci. 2019 May 1;16(5-6):46-49. PMID 31440402
- [Background] Martimbianco ALC, Porfirio GJ, Pacheco RL, Torloni MR, Riera R. Transcutaneous electrical nerve stimulation (TENS) for chronic neck pain. Cochrane Database Syst Rev. 2019 Dec 12;12(12):CD011927. doi: 10.1002/14651858.CD011927.pub2. PMID 31830313
- [Background] Reichstein L, Labrenz S, Ziegler D, Martin S. Effective treatment of symptomatic diabetic polyneuropathy by high-frequency external muscle stimulation. Diabetologia. 2005 May;48(5):824-8. doi: 10.1007/s00125-005-1728-0. Epub 2005 Apr 14. PMID 15830180
- [Background] DeSantana JM, Walsh DM, Vance C, Rakel BA, Sluka KA. Effectiveness of transcutaneous electrical nerve stimulation for treatment of hyperalgesia and pain. Curr Rheumatol Rep. 2008 Dec;10(6):492-9. doi: 10.1007/s11926-008-0080-z. PMID 19007541
- [Background] Doucet BM, Griffin L. High-versus low-frequency stimulation effects on fine motor control in chronic hemiplegia: a pilot study. Top Stroke Rehabil. 2013 Jul-Aug;20(4):299-307. doi: 10.1310/tsr2004-299. PMID 23893829
- [Background] Najafi B, Talal TK, Grewal GS, Menzies R, Armstrong DG, Lavery LA. Using Plantar Electrical Stimulation to Improve Postural Balance and Plantar Sensation Among Patients With Diabetic Peripheral Neuropathy: A Randomized Double Blinded Study. J Diabetes Sci Technol. 2017 Jul;11(4):693-701. doi: 10.1177/1932296817695338. Epub 2017 Feb 1. PMID 28627217
- [Background] Chandrasekaran S, Davis J, Bersch I, Goldberg G, Gorgey AS. Electrical stimulation and denervated muscles after spinal cord injury. Neural Regen Res. 2020 Aug;15(8):1397-1407. doi: 10.4103/1673-5374.274326. PMID 31997798
- [Background] Zehr EP, Collins DF, Chua R. Human interlimb reflexes evoked by electrical stimulation of cutaneous nerves innervating the hand and foot. Exp Brain Res. 2001 Oct;140(4):495-504. doi: 10.1007/s002210100857. PMID 11685403

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-29): https://cdn.clinicaltrials.gov/large-docs/58/NCT06421558/Prot_SAP_000.pdf